CLINICAL TRIAL: NCT07151573
Title: 5 Gode Vaner - En Randomisert Kontrollert Studie
Brief Title: Evaluating the Big Five Intervention in Norway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 911669
Record Dates: First submitted 2025-08-22; First posted 2025-09-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Depression
Keywords: Anxiety; Internet interventions; Big Five; DIgital Mental Health Intervention; Preventive interventions
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Three-armed randomized controlled study
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Big Five (Experimental)
  Interventions: Other: Big Five
- Gratitude (Active Comparator)
  Interventions: Other: Gratitude
- Waitlist (No Intervention): Waitlist during the intervention period, and receive Big Five on week 5.

INTERVENTIONS:
Other: Big Five — The intervention is self-guided and consists of a brief 14-page psychoeducation module that they are introduced to in the beginning of a 4-week intervention period (day 0). The module starts with a general introduction to mental health and Things you do action and how it promotes mental health. The final section presents the five core actions: 1) healthy thinking, 2) meaningful activities, 3) goals and plans, 4) healthy habits, and 5) social connections. Participants are advised to engage in the five daily actions throughout the intervention period. They are also encouraged to fill out a weekly planner and monitor their progress by keeping an overview of the number of daily activities in "My Week".The participants receive the module on a Sunday (Day 0). They receive text reminders Monday to Friday for four weeks, encouraging them to engage in the actions.
  Other Names: TYD
  Arms: Big Five
Other: Gratitude — The intervention is self-guided and consists of a brief 14-page psychoeducation module that they are introduced to in the beginning of a 4-week intervention period (day 0). The module starts with a general introduction to mental health and Gratitude and how it promotes mental health, followed by a short summary on the benefits of gratitude. The final section introduces practical strategies for cultivating gratitude by focusing on five key gratitude activities: 1) keeping a gratitude journal, 2) expressing gratitude to others, 3) finding gratitude in misfortune or difficult situations, 4) appreciating good things and 5) another perspective. The participants receive the module on a Sunday (Day 0). They receive text reminders Monday to Friday for four weeks, encouraging them to engage in the actions.
  Arms: Gratitude

SUMMARY:
This randomized controlled trial will evaluate the Norwegian adaptation of the Big Five intervention (Things You Do; TYD) for individuals with self-reported anxiety and/or depressive symptoms. The study will compare the Big Five intervention with a Gratitude intervention and a waitlist control. A total of 410 participants will be recruited online and randomized to one of three groups. Intervention groups will receive a brief module and daily SMS reminders (Monday-Friday for four weeks) encouraging engagement in either the five daily actions or gratitude practices. The primary aim is to replicate findings from the Australian trial by comparing TYD to a waitlist control. A secondary aim is to examine whether TYD yields better outcomes than the active Gratitude control. This study will provide evidence on the effectiveness and cross-cultural applicability of a low-cost, scalable intervention for improving mental health. Data from the study will also be used to evaluate the psychometric properties of the Norwegian translation of the Things You Do-15 instrument (TYD-15).

DETAILED DESCRIPTION:
Researchers in Australia have identified five central daily actions that are associated with mental health and may account for 37 % of the variance in anxiety and depressive symptoms: Healthy thinking, Meaningful Activities, Goals and Plans, Healthy Habits, and Social Connections. Conducting these actions more than three to four times a week may improve symptoms of anxiety and depression. Aim: The current study aims to replicate the findings from the Australian developers by adapting the intervention to a Norwegian context in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* PHQ or GAD cutoff 5 or above
* Residing in Norway and have a Norwegian national identity number
* 16 years or above

Exclusion Criteria:

* Reporting 2 or higher on PHQ item 9 (suicidality concerns)
* Do not comprehend Norwegian or English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder- 7 | At Screening
  the scale measures measure anxiety symptoms over the last two weeks. The questionnaire consists of seven items on a 4-point Likert Scale ranging from 0 (Not at all) to 3 (Nearly every day), giving a minimum score of 0 and maximum 21. Higher scores indicate more anxiety symptoms.
Patient Health Questionnaire - 2 | At pre, day 8, day 15, day 22, post, follow-up 3, 6, and 12 months
  The scale measures depressive symptoms symptoms over the last two weeks. The questionnaire consists of two items on a 4-point Likert Scale ranging from 0 (Not at all) to 3 (Nearly every day), giving a minimum score of 0 and maxiumum 6. Higher scores indicate more depressive symptoms.
Patient Health Questionnaire - 9 | At screening
  The scale measures depressive symptoms symptoms over the last two weeks. The questionnaire consists of nineitems on a 4-point Likert Scale ranging from 0 (Not at all) to 3 (Nearly every day), giving a minimum score of 0 and maximum 27. Higher scores indicate more depressive symptoms.
Generalized Anxiety Disorder - 2 | At pre, day 8, day 15, day 22, post, follow-up 3, 6, and 12 months
  The scale measures anxiety symptoms symptoms over the last two weeks. The questionnaire consists of two items on a 4-point Likert Scale ranging from 0 (Not at all) to 3 (Nearly every day), giving a minimum score of 0 and maxiumum 6. Higher scores indicate more anxiety symptoms.

SECONDARY OUTCOMES:
Satisfaction With Life Scale | From pre, peri intervention, post, and follow-up 3, 6 and 12 months
  The scale measure subjective well-being and life satisfaction. The questionnaire consists of five items on a 7-point Likert scale ranging from 1 (Strongly disagree) to 7 (Strongly agree), giving a minimum sum score of 5 and maximum 35. Higher scores indicate greater life satisfaction.

OTHER OUTCOMES:
Gratitude Questionnaire | From pre, peri intervention, post, and follow-up 3, 6 and 12 months
  The scale measure their experience of gratitude. The questionnaire consists of 6 items on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree), with two of the questions being reversed scored, giving a minimum sum score of 6 and a maximum score of 42. Higher scores indicate greater experience of gratitude.
Things You Do-15 Questionnaire | At screening, pre, peri intervention, post, and follow-up 3, 6 and 12 months
  TYD.15 measure their engagement in the daily actions that are associated with emotional wellbeing. The questionnaire comprises of 15 items on a scale from 0 to 4, giving a minimum sum score of 0 and maximum 60. Higher sum scores indicate greater engagement in daily actions.
Motivation for change in daily life - Questionnaire | day 8
  The scale measure their motivation and the importance of making changes in habits, readiness to change, and confidence in that they can make changes. The questionnaire consists of total 4 items on a scale from 1 to 10. Higher score on each item indicate greater motivation
Credibility | day 8, post
  Credibility is a 1-item assessment measuring whether they would recommend the intervention to a friend on a scale from 1 to 9. Higher score indicate greater credibility.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Research centre for digital mental health services, Bergen, Vestland
  - Research Centre For Digital Mental Health Services - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: When data collection ends
Access Criteria: IPD will be made available from PI on reasonable request and according to relevant Norwegian laws and regulations